CLINICAL TRIAL: NCT07058090
Title: Comparison of the Outcome of Treatment With Silymarin or N-Aceylcysteine in Patients Taking Anti-Tuberculous Drugs for Tuberculosis at a Tertiary Care Hospital , Karachi
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Liaquat National Hospital & Medical College (Other)
Responsible Party: Principal Investigator, Ariba SULTAN, Principal investigator, Liaquat National Hospital & Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1188-2025-LNH-ERC
Record Dates: First submitted 2025-06-26; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Drug Induced Liver Injury; Tuberculosis (TB)
Keywords: prevention of Antituberculous drugs induced liver injury
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury; Tuberculosis | interventions — Silymarin; Acetylcysteine; Rifampin; Ethambutol; Isoniazid; Protons; Pyrazinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group C (Active Comparator): patients taking antituberculous drugs only
  Interventions: Drug: Rifampicin (RMP) Ethambutol (E) Isoniazid (H) Pyrazinamid (Z)
- group A (Experimental): patients taking antituberculous drugs with silymarin
  Interventions: Drug: Silymarin 420 mg
- group B (Experimental): patients taking antituberculous drugs with N-acetylcysteine
  Interventions: Drug: N Acetyl Cysteine

INTERVENTIONS:
Drug: Silymarin 420 mg — silymarin group received silymarin 140mg thrice daily along with antituberculous drugs for 14 days
  Arms: group A
Drug: N Acetyl Cysteine — N- acetylcysteine group will receive N-acetylcysteine 900mg once daily with antituberculous drugs for 14 days
  Arms: group B
Drug: Rifampicin (RMP) Ethambutol (E) Isoniazid (H) Pyrazinamid (Z) — Antituberculous drugs only
  Arms: group C

SUMMARY:
OBJECTIVE : To compare the outcome of treatment with silymarin or N-acetyl cysteine in patients taking anti-tuberculous drugs for tuberculosis at Tertiary Care Hospital, Karachi.

SAMPLE SELECTION : Patients presenting with tuberculosis previously not on anti-tuberculous drugs, between 40-80 years of age, both genders will be included .Patients with history of alcohol use,Discontinuation of drug due to other adverse effects except hepatotoxicity ,Inadequate date of laboratory testing at baseline or 2 to 4 weeks after treatment initiation, Cases with human immunodeficiency virus (HIV) co-infection, viral hepatitis, or suspected mal absorption (e.g., gastrointestinal disease or diarrhea) ,Chronic liver disease, COPD, asthma, myocardial infarction, chronic kidney disease and stroke will be excluded

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with tuberculosis and previously not on any anti-tuberculous drugs, between 40-80 years of age
* either gender.

Exclusion Criteria:

* History of malignancy.
* Patients with history of seropositive, seronegative, connective tissue disorder or vasculitis, congestive cardiac failure.
* Patients with history of alcohol use.
* Discontinuation of drug due to other adverse effects except hepatotoxicity.
* Inadequate date of laboratory testing at baseline or 2 to 4 weeks after treatment initiation.
* Cases with human immunodeficiency virus (HIV) co-infection, viral hepatitis, or suspected mal absorption (e.g., gastrointestinal disease or diarrhea).
* Chronic liver disease, COPD, asthma, myocardial infarction, chronic kidney disease and stroke.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Anti-Tuberculous Drug induced Hepatotoxicity | 14 days
  Outcome will be assessed in patients developing Anti-tuberculous Drug-Induced Hepatotoxicity. Patients diagnosed with TB and started on a regimen based on isoniazid, rifampicin, pyrazinamide, and ethambutol will be labeled as having Anti-tuberculous Drug-Induced Hepatotoxicity using liver function tests. It will be labeled if any one of the following criteria is met:
  * Rise in alanine aminotransferase (ALT) more than or equal to a fivefold increase from the upper limit of normal (>37 IU/L)
  * Rise in alkaline phosphatase (ALP) more than or equal to twofold increase from the upper limit of normal (>147 IU/L).
  * An increase in alanine aminotransferase (ALT) to three or more times the upper normal limit (greater than 37 IU/L), accompanied by a simultaneous rise in bilirubin levels to more than twice the upper normal limit (exceeding 1.5 mg/dL), will be considered significant.

CONTACTS AND LOCATIONS:
Overall Officials: Ariba Sultan, Principal Investigator — Liaquat National Hospital & Medical College

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luangchosiri C, Thakkinstian A, Chitphuk S, Stitchantrakul W, Petraksa S, Sobhonslidsuk A. A double-blinded randomized controlled trial of silymarin for the prevention of antituberculosis drug-induced liver injury. BMC Complement Altern Med. 2015 Sep 23;15:334. doi: 10.1186/s12906-015-0861-7. PMID 26400476
- [Background] Ejigu DA, Abay SM. N-Acetyl Cysteine as an Adjunct in the Treatment of Tuberculosis. Tuberc Res Treat. 2020 Apr 30;2020:5907839. doi: 10.1155/2020/5907839. eCollection 2020. PMID 32411461
- [Background] Safe IP, Lacerda MVG, Printes VS, Praia Marins AF, Rebelo Rabelo AL, Costa AA, Tavares MA, Jesus JS, Souza AB, Beraldi-Magalhaes F, Neves CP, Monteiro WM, Sampaio VS, Amaral EP, Gomes RS, Andrade BB, Cordeiro-Santos M. Safety and efficacy of N-acetylcysteine in hospitalized patients with HIV-associated tuberculosis: An open-label, randomized, phase II trial (RIPENACTB Study). PLoS One. 2020 Jun 26;15(6):e0235381. doi: 10.1371/journal.pone.0235381. eCollection 2020. PMID 32589648
- [Background] Mahakalkar SM, Nagrale D, Gaur S, Urade C, Murhar B, Turankar A. N-acetylcysteine as an add-on to Directly Observed Therapy Short-I therapy in fresh pulmonary tuberculosis patients: A randomized, placebo-controlled, double-blinded study. Perspect Clin Res. 2017 Jul-Sep;8(3):132-136. doi: 10.4103/2229-3485.210450. PMID 28828308